CLINICAL TRIAL: NCT04477278
Title: Examining the Impact of Mindfulness on Patients' Experience of Osteopathic Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adam Hanley, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_00116896
Record Dates: First submitted 2020-07-13; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Pain; Satisfaction, Patient
MeSH Terms: conditions — Pain; Patient Satisfaction | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audio-Guided Mindfulness Intervention (Experimental): Brief, 8-minute, audio-guided mindfulness intervention delivered prior to osteopathic manipulation.
  Interventions: Behavioral: Mindfulness Meditation
- History of Osteopathy (Active Comparator): Brief, 8-minute, audio-guided history of osteopathy delivered prior to osteopathic manipulation.
  Interventions: Behavioral: History of Osteopathy

INTERVENTIONS:
Behavioral: Mindfulness Meditation — The mindfulness meditation recording consisted of instruction in focused attention on breath and body sensations and metacognitive monitoring and acceptance of discursive thoughts, negative emotions, and pain.
  Arms: Audio-Guided Mindfulness Intervention
Behavioral: History of Osteopathy — The history of osteopathy recording introduced patients to the founder of osteopathy, Andrew Taylor Still, and his philosophy of healing.
  Arms: History of Osteopathy

SUMMARY:
This is a single site, two-arm, parallel group pilot randomized controlled trial examining the effect of coupling a brief mindfulness-based intervention with an osteopathic manipulation session for pain patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for OMT at the Huntsman Cancer Institute

Exclusion Criteria:

* Altered mental status due to delirium, psychosis, or medication sedation as determined by treating clinician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity from immediately before session to immediately after | Immediately before and after the osteopathic manipulation session (i.e., 1 hour)
  Pain intensity was measured with individual items rated on a numeric rating scale (0-10). Higher scores indicate more pain.

SECONDARY OUTCOMES:
Change in Sensation Ratio (Pleasant/Unpleasant) from immediately before session to immediately after | Immediately before and after the osteopathic manipulation session (i.e., 1 hour)
  The sensation manikin is a digital human figure silhouette that is overlaid with a grid of 786 "sensation" pixels. Participants identify locations (i.e., grid pixels) on the manikin where they feel both pleasant and unpleasant sensations. Clicking once on any grid pixel turns that location blue, indicating a pleasant sensation. Clicking twice on any grid pixel turns that location red, indicating an unpleasant sensation. Each participant was instructed to color the entire area in which they were currently feeling sensation in their body. A clinically useful sensation ratio score is achieved by dividing the number of pleasant sensation pixels reported by the number of unpleasant sensation pixels reported. Higher scores indicate a larger pleasant sensation to unpleasant sensation ratio.
Patient Satisfaction | Immediately after the osteopathic manipulation session
  Session satisfaction was measured with an individual item ("I am satisfied with my treatment session.") rated on a numeric rating scale (0-10). Higher scores indicate greater satisfaction.
Change in Mindfulness of the Body from immediately before pre-session audio recording to immediately after | Immediately before and after the pre-session audio recording (i.e., 10 minutes)
  Mindfulness of the body was measured with an individual item ("I felt in contact with my body") from the State Mindfulness Scale (Tanay & Bernstein, 2013) rated on a numeric rating scale (0-10). Higher scores indicate more mindfulness of the body.
Change in Embodied Safety from immediately before pre-session audio recording to immediately after | Immediately before and after the pre-session audio recording (i.e., 10 minutes)
  Embodied safety was measured with an individual item ("I felt my body was a safe place."), from the Multidimensional Assessment of Interoceptive Awareness (Mehling et al., 2012) rated on a numeric rating scale (0-10). Higher scores indicate greater embodied safety.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available to qualified applicants upon receipt of worthy project proposal

REFERENCES:
- [Derived] Hanley AW, Wilson Zingg R, Smith B, Zappa M, White S, Davis A, Worts PR, Culjat C, Martorella G. Mindfulness in the Clinic Waiting Room May Decrease Pain: Results from Three Pilot Randomized Controlled Trials. J Integr Complement Med. 2024 Nov;30(11):1082-1091. doi: 10.1089/jicm.2024.0020. Epub 2024 May 17. PMID 38757714